CLINICAL TRIAL: NCT03621163
Title: Shade Evaluation for Clinical Color Change of Discolored Teeth Treated by Bleaching vs Laminate Veneers.
Brief Title: Copmere Between Bleaching and Laminate Veneers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hazim sherif ahmed, Dentist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DTB&V
Record Dates: First submitted 2018-07-29; First posted 2018-08-08 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Discoloration, Tooth
Keywords: bleaching agent
MeSH Terms: conditions — Tooth Discoloration | interventions — Bleaching Agents

STUDY DESIGN:
Intervention Model Description: split mouth randomized control, co-supervisor will write number for each member in each group (left side treatment A, right side treatment B or left side treatment B, right side treatment A) by indispensible pen on large white paper sheet. The sheet will be folded eight times and saved inside opaque well sealed envelope in which the inner content cannot be seen by naked eyes.
Who Masked: Outcomes Assessor
Masking Description: Single blinded (outcome assessor). Assessors supervisor and co-supervisor will be blinded to the assigned material. However the operator and patient can't be blinded due to the difference in preparation and shade of the ceramic materials and bleaching agent.
  * The assessors will assess all outcomes blinded to the material assigned for each patient.
  * Three spectrophotometer measurements will be recorded each time, with the active point of the instrument focused on the cervical third of each tooth, then mean color from three measurements will be calculated.
  * Digital photograph measures the color of teeth based on the Adobe Photoshop software. (Version 5.5).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bleaching agent (Experimental): intervention : bleaching agent ( Boost 40%)
  Interventions: Procedure: Bleaching agent ( BOOST 40%)
- laminate veneers (Active Comparator): laminate veneers ( monolithic lithium - silicate)
  Interventions: Procedure: laminate veneers(lithium-silicate)

INTERVENTIONS:
Procedure: Bleaching agent ( BOOST 40%) — Opalescence Boost 40% is a 40% hydrogen peroxide, medical power bleaching gel. The jet mix syringe ensures freshness for each application and precise dosing of the activator. One barrel contains a unique chemical activation with sodium fluoride and potassium nitrate, which have been demonstrated to reduce caries susceptibility, lower sensitivity, and improve enamel micro-hardness. The other barrel contains the concentrated hydrogen peroxide. When mixed, Opalescence Boost results in a 1.1% fluoride and 3% potassium nitrate concentration.
  Arms: bleaching agent
Procedure: laminate veneers(lithium-silicate) — A lithium-silicate glass ceramic is newly introduced to the market. After crystallization, it demonstrates an ideal combination of strength, aesthetics and translucency that mirrors the vitality of natural teeth for fabrication of full anatomic anterior and posterior crowns. It differentiated from other ceramics by its high chipping resistance, due to their monolithic composition and average flexural strength of 385 MPa. Also Milling Block has good wear resistance due to the high content of ultra-fine nano-meter size crystalline structure. Lithium-silicates ceramic blocks are available in the commonly used VITA Classical and Chromascop Bleach shades.
  Arms: laminate veneers

SUMMARY:
The present study is aimed to evaluation of shade for clinical color change of discolored teeth treated by bleaching vs laminate veneers.

DETAILED DESCRIPTION:
Dental aesthetics, including tooth color, is of great importance for majority of the people and any discoloration or staining can affect their quality of life negatively1,2. In the UK it has been reported that 28% of grownups are dissatisfied with the appearance of their teeth and in the USA that 34% of grownups population are dissatisfied with their current tooth color. Moreover, in a survey of 3215 subjects from the UK 50% have admitted that they had some kind of tooth discoloration3,4.

Tooth bleaching has become one of the most popular aesthetic dental treatments. Because tooth bleaching is an effective, non-invasive procedure for the change of tooth discoloration, it is the best of treatment options for improving teeth color 5.

Ceramic restorations with excellent biocompatibility are widely used to achieve highly aesthetic characteristics in ﬁxed prosthodontics6. Porcelain laminate veneers have become a popular method of treated tooth discoloration. But are expensive, brittle and difficult to repair7.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in this clinical trial :

  * Men and women between 15and 40 years of age.
  * Had good general and oral health.
  * The participants needed to have six vital maxillary or mandibular anterior teeth without caries lesions or restorations.
  * The maxillary canine was shade A3 or darker as judged by comparison with a shade guide (VITA Classical Shade Guide or Spectrophotometer measurement ).

Exclusion Criteria:

* Participants were excluded from the study

  * If they presented with anterior restorations; had bruxism habits.
  * Were pregnant/lactating; presented with non vital tooth discoloration.
  * were taking any drug with anti-inflammatory, analgesic, or antioxidant effect; or presented with recession and dentin exposure

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1 (Estimated)
Dates: Start 2018-12-05 (Estimated); Primary Completion 2019-09-05 (Estimated); Study Completion 2019-12-20 (Estimated)

PRIMARY OUTCOMES:
Color change. | 1-4 weeks
  measures the change of color before and after intervention by Easy Shade Spectrophotometry

SECONDARY OUTCOMES:
Corresponding color with comparator. | 1-4 weeks
  by Digital photographs

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gupta SK, Saxena P. Evaluation of patient satisfaction after non-vital bleaching in traumatized discolored intact anterior teeth. Dent Traumatol. 2014 Oct;30(5):396-399. doi: 10.1111/edt.12109. Epub 2014 Apr 10. PMID 24720860
- [Background] Gerlach RW, Zhou X. Clinical trial comparing two daytime hydrogen-peroxide professional vital-bleaching systems. Compend Contin Educ Dent. 2004 Aug;25(8 Suppl 2):33-40. PMID 15645893
- [Background] Almeida LC, Riehl H, Santos PH, Sundfeld ML, Briso AL. Clinical evaluation of the effectiveness of different bleaching therapies in vital teeth. Int J Periodontics Restorative Dent. 2012 Jun;32(3):303-9. PMID 22408775
- [Background] Mountouris G, Mantzavinos Z, Michou H. [Discolorations: a new method of bleaching discolored vital teeth. (Preliminary study)]. Odontostomatol Proodos. 1990 Jun;44(3):195-206. Greek, Modern. PMID 2130332
- [Background] Marson FC, Sensi LG, Vieira LC, Araujo E. Clinical evaluation of in-office dental bleaching treatments with and without the use of light-activation sources. Oper Dent. 2008 Jan-Feb;33(1):15-22. doi: 10.2341/07-57. PMID 18335728
- [Background] Alomari Q, El Daraa E. A randomized clinical trial of in-office dental bleaching with or without light activation. J Contemp Dent Pract. 2010 Jan 1;11(1):E017-24. PMID 20098962